CLINICAL TRIAL: NCT04649229
Title: Mechanisms Underlying Hypotensive Response to ARB/NEP Inhibition - Aim 3
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Nancy Brown, Professor of Internal Medicine, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2000028712
Record Dates: First submitted 2020-11-12; First posted 2020-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; p-Aminohippuric Acid; Iohexol; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- placebo, aprepitant, placebo, aprepitant (Experimental): After a 48-hr washout, participants in this arm will be given LCZ696 50 mg and placebo (vehicle). After a 96-hr washout period, subjects will be given LCZ696 50 mg and aprepitant. Participants will then undergo uptitration of LCZ696 over seven weeks. On the 7th and 10th days of the 200 mg bid or highest tolerated dose of LCZ696, participants in this arm will receive placebo and aprepitant, respectively.
  Interventions: Drug: LCZ 696; Drug: Placebo; Drug: Para-aminohippurate; Drug: Iohexol; Drug: Aprepitant
- placebo, aprepitant, aprepitant, placebo (Experimental): After a 48-hr washout, participants in this arm will be given LCZ696 50 mg and placebo (vehicle). After a 96-hr washout period, subjects will be given LCZ696 50 mg and aprepitant. Participants will then undergo uptitration of LCZ696 over seven weeks. On the 7th and 10th days of the 200 mg bid or highest tolerated dose of LCZ696, participants in this arm will receive aprepitant and placebo, respectively.
  Interventions: Drug: LCZ 696; Drug: Placebo; Drug: Para-aminohippurate; Drug: Iohexol; Drug: Aprepitant
- aprepitant, placebo, placebo, aprepitant (Experimental): After a 48-hr washout, participants in this arm will be given LCZ696 50 mg and aprepitant. After a 96-hr washout period, subjects will be given LCZ696 50 mg and placebo. Participants will then undergo uptitration of LCZ696 over seven weeks. On the 7th and 10th days of the 200 mg bid or highest tolerated dose of LCZ696, participants in this arm will receive placebo and aprepitant, respectively.
  Interventions: Drug: LCZ 696; Drug: Placebo; Drug: Para-aminohippurate; Drug: Iohexol; Drug: Aprepitant
- aprepitant, placebo, aprepitant, placebo (Experimental): After a 48-hr washout, participants in this arm will be given LCZ696 50 mg and aprepitant. After a 96-hr washout period, subjects will be given LCZ696 50 mg and placebo. Participants will then undergo uptitration of LCZ696 over seven weeks. On the 7th and 10th days of the 200 mg bid or highest tolerated dose of LCZ696, participants in this arm will receive aprepitant and placebo, respectively.
  Interventions: Drug: LCZ 696; Drug: Placebo; Drug: Para-aminohippurate; Drug: Iohexol; Drug: Aprepitant

INTERVENTIONS:
Drug: LCZ 696 — Treatment with LCZ696 is unblinded in this study. After the two acute study days, subjects will be provided LCZ696 50 mg bid for two weeks. At the end of those two weeks subjects will report to the Clinical Research Center (CRC) for a dose escalation visit. If their tolerance, blood pressure, potassium, and eGFR meet escalation criteria they will be given LCZ696 100 mg bid for three weeks. (If they do not meet escalation criteria they will be continued on LCZ696 50 mg bid.) After three weeks, they will return to the CRC for the next escalation visit. If they meet criteria for escalation they will be given LCZ 200 mg bid for ten days. (If they do not meet escalation criteria they will be continued on the highest tolerated dose).
  Other Names: Entresto
Drug: Placebo — Placebo or aprepitant 120 mg will be given orally on study days 1 and 2 and again on study days 3 and 4
Drug: Para-aminohippurate — Para-aminohippurate (PAH) will be given at a dose of 8 mg/kg loading dose followed by a 12 mg/min steady-state infusion during each study day.
Drug: Iohexol — Iohexol will be given as 5 mL of iohexol solution (3.235 g iohexol) intravenously on each study day.
Drug: Aprepitant — Placebo or aprepitant 120 mg will be given orally on study days 1 and 2 and again on study days 3 and 4

SUMMARY:
This is a double-blind, randomized, two x two crossover (aprepitant vs placebo) during both initiation of Entresto, LCZ696, (50 mg dose) and at steady-state of Entresto (200 mg bid dose or the highest tolerated dose).

DETAILED DESCRIPTION:
LCZ696, a molecular complex of the angiotensin receptor blocker (ARB) valsartan with an inhibitor of neprilysin (NEP, neutral endopeptidase-24.11) sacubitril improved mortality compared to enalapril in patients with heart failure (HF), reduced ejection fraction (EF), and increased brain natriuretic peptide (BNP) or N-terminal pro-BNP (NT-proBNP) in the PARADIGM-HF trial. The PIONEER-HF study demonstrated the efficacy of LCZ696 in preventing rehospitalization in patients with acutely decompensated HF.

LCZ696 has been underutilized in heart failure, in part due to concerns about hypotension. NEP degrades several vasodilator peptides including bradykinin, substance P and brain-type natriuretic peptide. Decreased degradation of endogenous substance P could contribute to hypotension at initiation of LCZ696 through vasodilation or through increased natriuresis and diuresis. Antagonism of the NK1 receptor using aprepitant would be expected to prevent this effect.

Objectives

The main objectives of this mechanistic randomized, double-blind, crossover-design study are:

The primary objective is to test the hypothesis that endogenous substance P contributes to effects of ARB/NEP inhibition on blood pressure, natriuresis, and diuresis at initiation.

The secondary objective is to test the hypothesis that endogenous substance P contributes to effects of ARB/NEP inhibition on blood pressure, natriuresis, and diuresis after up-titration.

Eighty (80) subjects with stable heart failure who meet all inclusion/exclusion criteria will be enrolled. Subjects who qualify will collect their urine for 24 hours before each study day for measurement of volume, sodium and potassium. At the start of the study, they will stop their regular angiotensin-converting enzyme (ACE) inhibitor or ARB. After a 48-hour washout, they will undergo a study day in which they are given a single dose of 50 mg LCZ696. They will also receive either the NK1 receptor antagonist aprepitant or placebo vehicle in random order (double-blind). After a 96-hour washout, they will repeat the study day and receive a single dose of 50 mg LCZ696 and the opposite study drug (aprepitant or placebo). After completion of the two acute study days, subjects will take LCZ696 50 mg bid for two weeks, followed by LCZ696 100 mg bid for three weeks, and then LCZ696 200 mg bid, following the conservative up-titration protocol from the TITRATION study. Criteria for continuing up-titration appears in the full study protocol. On the 7th and 10th day of the 200 mg bid or highest tolerated dose, subjects will again undergo two more study days three days apart in which they are randomized to receive either aprepitant or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Black and white men and women
2. Stable patients with a reduced ejection fraction (EF)

   1. EF ≤55%, and
   2. history of symptoms of New York Heart Association (NYHA) class I, II, or III heart failure (HF)
   3. stable clinical symptoms including no hospitalizations for the last three months, or one month if hospitalized only once for initial diagnosis of HF
   4. who are not already taking LCZ696
3. treatment with a stable dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) and with a beta blocker (unless contraindicated or not tolerated) for at least four weeks
4. for patients with NYHA Class II or III HF and EF ≤35%, treatment with a stable dose of an mineralocorticoid receptor (MR) antagonist for at least four weeks, unless not possible due to renal function or adverse reaction
5. For female subjects, the following conditions must be met:

   1. postmenopausal status for at least one year
   2. status post-surgical sterilization
   3. or if childbearing potential, utilization of barrier methods of birth control or an oral contraceptive and willingness to undergo urine β-HCG testing on every study day
6. Age 18 years of age or older

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACEi, ARBs, or neutral endopeptidase inhibitor (NEPi), as well as known or suspected contraindications to the study drugs
2. History of angioedema
3. History of decompensated HF within the last 3 months (exacerbation of chronic HF manifested by signs and symptoms that required intravenous therapy or hospitalization) or one month if hospitalized only once for initial diagnosis of HF
4. History of heart transplant or on a transplant list or with left ventricular assistance device
5. Symptomatic hypotension and/or a systolic blood pressure (SBP)<100 mmHg at screening or <95 mmHg during the study
6. Serum potassium >5.2 mmol/L at screening or during the study
7. Impaired renal function (eGFR of <30mL/min/1.73 m2) as determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine (Scr) is expressed in mg/dL and age in years:

   a. eGFR (mL/min/1.73 m2)=175 • Scr-1.154 • age-0.203 • (1.212 if Black) • (0.742 if female)
8. Acute coronary syndrome, cardiac, carotid, or other major cardiovascular surgery, percutaneous coronary intervention, or carotid angioplasty within six months prior to screening
9. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within six months of screening
10. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack with clinically significant residual deficits
11. History of ventricular arrhythmia with syncopal episodes
12. Symptomatic bradycardia or second- or third-degree atrioventricular block without a pacemaker
13. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular (LV) dilatation
14. Presence of other hemodynamically significant obstructive lesions of the LV outflow tract, including aortic and subaortic stenosis
15. Type 1 diabetes
16. Poorly controlled type 2 diabetes mellitus (T2DM), defined as a HgbA1c >9%
17. In T2DM, dipeptidyl peptidase-4 inhibitor use for one month prior to enrollment will be excluded due to possible interaction with LCZ696
18. Hematocrit <35%
19. Breast feeding and pregnancy
20. History or presence of immunological or hematological disorders
21. History of malignancy not felt to be cured, except non-melanoma skin cancer
22. Diagnosis of asthma requiring use of inhaled beta agonist more than once a week
23. History of hypersensitivity reaction to contrast
24. Clinically significant gastrointestinal impairment that could interfere with drug absorption
25. History of pancreatitis or known pancreatic lesions
26. Impaired hepatic function with evidence of advanced fibrosis or cirrhosis [stable aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) trend if >3.0 x upper limit of normal range as deemed of minimal clinical relevance by the investigators]
27. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal anti-inflammatory drugs
28. Treatment with greater than 5 mg of prednisone or equivalent dose of chronic systemic glucocorticoid therapy within the last year or recent (within 6 weeks of first study day) treatment with burst dosed glucocorticoid therapy
29. Treatment with lithium salts
30. History of alcohol or drug abuse
31. Treatment with any investigational drug in the one month preceding the study
32. Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
33. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) | Over six hours on each of the four study days
  Mean arterial pressure (MAP) will be measured before and after administration of LCZ696 on each of the four study days
Urine sodium excretion | Total urine output from drug administration to six hours following drug administration
  Urine sodium excretion will be measured for six hours following administration of LCZ696 on each of the four study days.

SECONDARY OUTCOMES:
Heart rate | Over six hours on each of four study days
  Heart rate (HR) will be measured before and after LCZ696 on each of the four study days
Urine volume | Over six hours on each of four study days
  Urine volume will be measured for six hours following LCZ696 on each of the four study days.
Renal plasma flow | Over six hours on each of four study days
  Renal plasma flow (RPF) will be calculated from para-aminohippurate clearance prior to and following LCZ696.
Glomerular filtration rate | Over six hours on each of four study days
  Glomerular filtration rate (GFR) will be calculated from the clearance of iohexol prior to and following LCZ66 on each of the four study days
Urine albumin-to-creatinine ratio | Over six hours on each of four study days
  Urine albumin-to-creatinine ratio (UACR) will be calculated before and after LCZ696 on each of the four study days.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Brown, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601
- [Background] Senni M, McMurray JJ, Wachter R, McIntyre HF, Reyes A, Majercak I, Andreka P, Shehova-Yankova N, Anand I, Yilmaz MB, Gogia H, Martinez-Selles M, Fischer S, Zilahi Z, Cosmi F, Gelev V, Galve E, Gomez-Doblas JJ, Nociar J, Radomska M, Sokolova B, Volterrani M, Sarkar A, Reimund B, Chen F, Charney A. Initiating sacubitril/valsartan (LCZ696) in heart failure: results of TITRATION, a double-blind, randomized comparison of two uptitration regimens. Eur J Heart Fail. 2016 Sep;18(9):1193-202. doi: 10.1002/ejhf.548. Epub 2016 May 12. PMID 27170530